CLINICAL TRIAL: NCT02982941
Title: A Phase 1, Open-label, Dose Escalation Study of MGA271 in Pediatric Patients With B7-H3-Expressing Relapsed or Refractory Solid Tumors
Brief Title: Enoblituzumab (MGA271) in Children With B7-H3-expressing Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-04
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; Ewing Sarcoma; Wilms Tumor; Desmoplastic Small Round Cell Tumor
Keywords: Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; Ewing Sarcoma; Wilms Tumor; Desmoplastic Small Round Cell Tumor; pediatric
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; Sarcoma, Ewing; Wilms Tumor; Desmoplastic Small Round Cell Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation & Cohort Expansion (Experimental): enoblituzumab administered IV weekly
  Interventions: Drug: Enoblituzumab

INTERVENTIONS:
Drug: Enoblituzumab — enoblituzumab administered IV weekly for up to 96 weeks
  Other Names: MGA271

SUMMARY:
This study is a Phase 1, open-label, dose escalation and cohort expansion trial designed to characterize the safety, tolerability, PK, PD, immunogenicity and preliminary antitumor activity of enoblituzumab administered IV on a weekly schedule for up to 96 doses (approximately 2 years) in children and young adults with B7-H3-expressing relapsed or refractory malignant solid tumors.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, dose escalation and cohort expansion trial designed to characterize the safety, tolerability, PK, PD, immunogenicity and preliminary antitumor activity of enoblituzumab administered IV on a weekly schedule for up to 96 doses (approximately 2 years) in children and young adults with B7-H3-expressing relapsed or refractory malignant solid tumors.

The study consists of a Dose Escalation Phase to determine the MTD (or MAD) of enoblituzumab followed by a Cohort Expansion Phase to further define the safety and initial antitumor activity of enoblituzumab. In the cohort expansion phase, 5 cohorts of 10 patients each will be enrolled to further evaluate the safety and potential efficacy of enoblituzumab administered at the MTD/MAD in patients with:1) neuroblastoma - measurable disease, 2) neuroblastoma - non-measurable disease, 3) rhabdomyosarcoma, 4) osteosarcoma, and 5) Ewing's sarcoma, Wilms' tumor, desmoplastic small round cell tumors, or malignant solid tumors of any other histology that test positive for B7-H3.

All tumor evaluations will be carried out by both Response Evaluation Criteria in Solid Tumors (RECIST) and immune-related response criteria (irRC). Disease assessment in patients with neuroblastoma will use neuroblastoma overall response criteria.

ELIGIBILITY:
General Inclusion Criteria:

* Age at treatment 1 to 35 years.
* Relapsed or refractory malignant solid tumors of any histology for which no standard curative therapy is available (escalation phase).
* Histologically proven: neuroblastoma, rhabdomyosarcoma, osteosarcoma, Ewing's sarcoma/ primitive neuroectodermal tumor, Wilms tumor, desmoplastic small round cell tumor or malignant solid tumors of any other histology that test positive for B7-H3 .
* Must have malignant solid tumors that demonstrate B7-H3 expression at 2+ or greater levels on the membranous surface of at least 10% of tumor cells or ≥ 25% of tumor vasculature by IHC.
* With the exception of patients with non-measurable neuroblastoma patients must have measurable disease as per RECIST 1.1
* Karnofsky (patients ≥ 16 years)/Lansky (patients < 16 years) index ≥ 70.
* Acceptable laboratory parameters and adequate organ reserve.

Exclusion Criteria:

* Patients are to be excluded from the study if they have any of the following:
* Patients with a history of symptomatic central nervous system (CNS) unless they have been treated and are asymptomatic.
* Patients with any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic treatment within the past 2 years, and patients with a history of Grave's disease that are now euthyroid clinically and by laboratory testing.
* History of prior allogeneic bone marrow/stem-cell or solid organ transplantation.
* Patients receiving autologous stem cell transplantation must wait 8 weeks before initiation of study drug administration.
* Treatment with systemic chemotherapy or investigational therapy within 4 weeks of first study drug administration; other agents (e.g., biologics) within 2 weeks; radiation within 2 weeks; patients receiving 131I-MIBG therapy must wait 6 weeks prior to the initiation of study drug administration; corticosteroids (≥ 0.2 mg/kg/day prednisone or equivalent) or other immune suppressive drugs within the 2 weeks prior to the initiation of study drug administration.
* History of clinically significant cardiovascular disease
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug.
* Known positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome.
* Known history of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction.
* Second primary invasive malignancy that has not been in remission for greater than 2 years.
* History of severe trauma or major surgery within 4 weeks prior to the initiation of study drug administration.
* Known hypersensitivity to recombinant proteins, polysorbate 80 or any excipient contained in the drug formulation for enoblituzumab
* Patients in Canada may not have a history or evidence of latent or active tuberculosis infection.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12; Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of enoblituzumab. | Time of first dose through end of treatment (up to 2 years)
  Adverse events, SAEs, incidence of treatment-emergent AE

SECONDARY OUTCOMES:
Peak plasma concentration | Time of first dose through end of treatment (up to 96 weeks)
  PK of enoblituzumab
Number of participants that develop anti-drug antibodies | Time of first dose through end of treatment (up to 96 weeks)
  Proportion of patients who develop anti-MGA271 antibodies, immunogenicity
Antitumor activity of enoblituzumab | Time of first dose through end of treatment (up to 96 weeks)
  Anti-tumor activity of enoblituzumab using conventional RECIST 1.1 and immune related RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital, Stanford, Palo Alto, California
  - National Cancer Institute, Center for Cancer Research, Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - University of Wisconsin, American Family Children's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No